CLINICAL TRIAL: NCT01360034
Title: Nifedipine vs. Indomethacin in the Treatment of Preterm Labour and Short Cervix. A Randomized, Controlled Trial.
Brief Title: Nifedipine Versus Indomethacin in the Treatment of Preterm Labour
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Saint Thomas Hospital, Panama (Other)
Responsible Party: Principal Investigator, Osvaldo A. Reyes T., MD, Saint Thomas Hospital, Panama
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MHST2011-04
Record Dates: First submitted 2011-05-20; First posted 2011-05-25 (Estimated); Last update posted 2015-01-05 (Estimated); Status verified 2015-01

CONDITIONS: Obstetric Labor, Premature
Keywords: Obstetric labor, premature; Short cervix; Nifedipine; Indomethacin
MeSH Terms: conditions — Obstetric Labor, Premature | interventions — Nifedipine; Indomethacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nifedipine (Experimental): 108 patients will receive nifedipine as tocolytic for 48 hours.
  Interventions: Drug: Nifedipine
- Indomethacin (Experimental): 108 patients will receive indomethacin as tocolytic for 48 hours.
  Interventions: Drug: Indomethacin

INTERVENTIONS:
Drug: Nifedipine — Nifedipine: 20 mg as a single dose upon admission and then 10 mg vo every 8 hours for 48 hours.
  Arms: Nifedipine
Drug: Indomethacin — Indomethacin: 50 mg vo as a single dose upon admission and then 25 mg vo every 6 hours for 48 hours.
  Arms: Indomethacin

SUMMARY:
The purpose of this study was to compare the effectiveness of nifedipine versus indomethacin as tocolytic for the treatment of preterm labour with short cervix (< 2.5cms).

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women between 24 and 34 weeks of gestation.
* Cervical length (determined by transvaginal ultrasound) of 2.5 cms or less

Exclusion Criteria:

* All contraindications for tocolysis (fetal distress, abruptio placenta).
* Multiple pregnancy.
* All contraindications for the use of any of the two drugs (indomethacin or nifedipine).

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2015-12; Primary Completion 2016-05 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Reduction of preterm birth (before 48 hours, allowing use of corticosteroids). | 36 months

SECONDARY OUTCOMES:
Reduction of preterm labour (before 35 weeks). | 48 months
Adverse effects | 48 months
  To determine the frequency of maternal adverse effects related to the use of both drugs (nifedipine and indomethacin). These include the development of any type of rash, nausea, weakness/hypotension, headache, dyspepsy or bleeding disorders of any kind.

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Espinosa, Resident, Principal Investigator — Saint Thomas Hospital, Panama; Osvaldo Reyes, MD, Principal Investigator — Saint Thomas Hospital, Panama
Locations (1):
- Saint Thomas Hospital, Panama City, Provincia de Panamá, Panama

REFERENCES:
- [Derived] Wilson A, Hodgetts-Morton VA, Marson EJ, Markland AD, Larkai E, Papadopoulou A, Coomarasamy A, Tobias A, Chou D, Oladapo OT, Price MJ, Morris K, Gallos ID. Tocolytics for delaying preterm birth: a network meta-analysis (0924). Cochrane Database Syst Rev. 2022 Aug 10;8(8):CD014978. doi: 10.1002/14651858.CD014978.pub2. PMID 35947046